CLINICAL TRIAL: NCT01742702
Title: Non-Invasive HaemoDYNAMICs in Primary and Secondary Hypertension: the DYNAMIC-study
Brief Title: HaemoDYNAMICs in Primary and Secondary Hypertension
Acronym: DYNAMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tampere University (Other)
Collaborators: Finnish Foundation for Cardiovascular Research (Other); Paavo Nurmi Foundation (Unknown); Sigrid Jusélius Foundation (Other); Finnish Cultural Foundation (Other); Tampere Tuberculosis Foundation (Other); Medical Research Fund of the Tampere University Hospital, Finland (Other); Aarne Koskelo Foundation (Other); Finnish Medical Foundation (Network); Finnish Kidney Foundation (Unknown); Päivikki and Sakari Sohlberg Foundation, Finland (Other)
Responsible Party: Principal Investigator, Ilkka Pörsti, MD, MD, PhD, Professor of Internal Medicine, Tampere University
Other Study IDs: R06086M; 2006-002065-39 (EudraCT Number); 2009-014542-29 (EudraCT Number); R07110M (Other: Ethics Committee of Pirkanmaa Hospital District); R07053M (Other: Ethics Committee of Pirkanmaa Hospital District); R08012 (Other: Ethics Committee of Pirkanmaa Hospital District); R09103M (Other: Ethics Committee of Pirkanmaa Hospital District); R10056 (Other: Ethics Committee of Pirkanmaa Hospital District); R06086M (Other: Ethics Committee of Pirkanmaa Hospital District); R21094 (Other: Ethics Committee of Pirkanmaa Hospital District)
Record Dates: First submitted 2012-11-29; First posted 2012-12-05 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Primary Hypertension; Secondary Hypertension; Aortic Stenosis; Renal Insufficiency
Keywords: Blood pressure; Hypertension; Arterial stiffness; Cardiac output; Vascular resistance; Pulse wave reflection; Head-up tilt
MeSH Terms: conditions — Essential Hypertension; Aortic Valve Stenosis; Renal Insufficiency; Hypertension | interventions — Nitroglycerin; Albuterol; halofantrine; Arginine; Glycyrrhiza glabra extract; Glycyrrhizic Acid; Bisoprolol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, serum, urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- DYNAMIC (ongoing): Subjects with primary or secondary hypertension and normotensive control subjects. In addition haemodynamic recordings to 50 subjects suffering from chronic fatigue syndrome will be performed.
- AERO-DYNAMIC (recordings completed): Subjects who had voluntarily decided to participate in a professionally coached marathon school (Varala Sports Institute, Tampere) were given the chance for haemodynamic recordings before, during and after the training protocol.
  Interventions: Drug: Nitroglycerin 0.25 mg (single dose, no longer given since January 2017); Drug: Salbutamol 400 µg (single dose, no longer given since January 2017)
- Liquorice (recordings completed): Normotensive subjects, daily liquorice ingestion (daily glycyrrhizin dose 290-370 mg) for 2 weeks, haemodynamic measurements before and after the intervention.
  Interventions: Drug: Nitroglycerin 0.25 mg (single dose, no longer given since January 2017); Drug: Salbutamol 400 µg (single dose, no longer given since January 2017); Dietary Supplement: Liquorice (2 weeks, glycyrrhizin 290-370 mg daily, no longer given since 2012)
- Milk polypeptides (recordings completed): Daily ingestion of yoghurt containing small milk casein-derived polypeptides for 12 weeks versus placebo yoghurt.
  Interventions: Dietary Supplement: Small milk casein-derived polypeptides (12 weeks daily, recordings completed 2011)
- Bisoprolol (recordings completed): Hypertensive subjects, bisoprolol 5 mg once daily versus placebo in a double-blind, cross-over protocol.
  Interventions: Drug: Nitroglycerin 0.25 mg (single dose, no longer given since January 2017); Drug: Salbutamol 400 µg (single dose, no longer given since January 2017); Drug: Bisoprolol (5 mg daily for 3 weeks, recordings completed 2011)
- Aortic stenosis (ongoing): Subjects with aortic stenosis confirmed by echocardiography
- Methodological (recordings completed): 35 normotensive subjects who received research drugs (nitroglycerin, salbutamol, placebo resoriblet, placebo inhalation, L-arginine infusion, saline infusion) in a placebo-controlled, double-blinded manner
  Interventions: Drug: Nitroglycerin 0.25 mg (single dose, no longer given since January 2017); Drug: Salbutamol 400 µg (single dose, no longer given since January 2017); Drug: L-arginine (10 min infusion, no longer given since January 2017)
- Participants of Ironman Triathlon: Altogether 80 athletes participating in a full length Ironman competition. Non-invasive recordingds are performed under normal conditions during the training period and after completion of a full-length Ironman competition.

INTERVENTIONS:
Drug: Nitroglycerin 0.25 mg (single dose, no longer given since January 2017) — From the beginning of the study until the end of year 2016 a single dose of sublingual nitroglycerin was given to examine the associated acute haemodynamic effects (recordings completed).
  Other Names: Nitro resoriblet, Orion Pharma, Espoo, Finland
  Groups: AERO-DYNAMIC (recordings completed); Bisoprolol (recordings completed); Liquorice (recordings completed); Methodological (recordings completed)
Drug: Salbutamol 400 µg (single dose, no longer given since January 2017) — From the beginning of the study until the end of year 2016 a 400 µg dose of inhaled salbutamol was given to examine the associated acute haemodynamic effects (recordings completed).
  Other Names: Ventoline, GlaxoSmithKline, Uxbridge, Middlesex, UK
  Groups: AERO-DYNAMIC (recordings completed); Bisoprolol (recordings completed); Liquorice (recordings completed); Methodological (recordings completed)
Drug: L-arginine (10 min infusion, no longer given since January 2017) — From the beginning of the study until the end of year 2016 L-arginine infusion 10 mg/kg/min could be given for 10 minutes to examine acute haemodynamic effects (recordings completed).
  Other Names: L-arginine HCl 20 mg ml/l, B. Braun Ag, Melsungen, Germany
  Groups: Methodological (recordings completed)
Dietary Supplement: Liquorice (2 weeks, glycyrrhizin 290-370 mg daily, no longer given since 2012) — Daily liquorice intake (daily glycyrrhizin dose 290-370 mg) for two weeks, measurements before and after intervention (recordings completed).
  Other Names: Halva liquorice (TM), Kouvola liquorice (TM)
  Groups: Liquorice (recordings completed)
Dietary Supplement: Small milk casein-derived polypeptides (12 weeks daily, recordings completed 2011) — Daily intake of yoghurt containing small milk casein-derived polypeptides (12 weeks) and placebo yoghurt (12 weeks), measurements before and after intervention (recordings completed 2011).
  Other Names: Valio (TM) evolus yoghurt
  Groups: Milk polypeptides (recordings completed)
Drug: Bisoprolol (5 mg daily for 3 weeks, recordings completed 2011) — Bisoprolol 5 mg daily for 3 weeks and placebo tablet daily for 3 weeks, double-blind, randomized, placebo-controlled cross-over protocol. Measurements before and after interventions (recordings completed 2011).
  Other Names: Emconcor 5 mg, Merck KGaA, Darmstadt, Germany
  Groups: Bisoprolol (recordings completed)

SUMMARY:
The primary aim of the present study was to examine the haemodynamic changes in primary hypertension and secondary hypertension (renal diseases, endocrine diseases, obesity-associated hypertension) with a non-invasive haemodynamic measurement protocol utilizing radial pulse wave analysis and whole-body impedance cardiography in both supine position and during head-up tilt. For comparison, haemodynamics of subjects with chronic fatigue syndrome will also be recorded.

DETAILED DESCRIPTION:
Elevated blood pressure (BP) and related cardiovascular complications are the leading causes of morbidity and mortality in the modern world. In routine clinical practice, the haemodynamic status is commonly assessed by measuring heart rate and blood pressure at rest, which provides only limited information about functional haemodynamic status. In addition, the haemodynamic changes resulting in similar elevations of BP may differ substantially between patients and disorders.

Therefore, we investigated the haemodynamic changes in primary and secondary hypertension and in the control subjects with non-invasive radial pulse wave analysis and whole-body impedance cardiography. The method includes the determination of volume status using bioimpedance spectroscopy, determination of peripheral and central BP, cardiac function, vascular resistance, arterial compliance and indices of pulse wave reflection. Besides the measurements performed in the supine position, passive orthostatic challenge is included in the protocol to assess the upright functional haemodynamic status.

The repeatability and reproducibility of the protocol was first examined with a double-blind, randomized protocol in 35 subjects (methodological study group), and after that the administration of research drugs has been open-label. The effects of single doses of two largely endothelium-dependent agents, inhaled salbutamol and intravenous L-arginine, and one endothelium-independent agent, sublingual nitroglycerin, were investigated. However, challenges with the acute dosing of all medical compounds was terminated at the end of December 2016. Thereafter, the measurement protocol has included supine and upright recordings on the tilt-table, followed by supine measurements during paced breathing (15 breaths per minute for 5 minutes, 6 breaths per minute for 5 minutes) that modulate the autonomic nervous tone.

The study population has consisted of subgroups described below. The study protocol of each subgroup has been approved by the ethics committee of the Pirkanmaa Hospital District (Ethics committee ID's above), and the administration of research drugs has also been approved by the Finnish Agency for Medicines (EudraCT-numbers above).

ELIGIBILITY:
Inclusion Criteria:

* Independent, community-dwelling adults
* Hypertensive subjects (primary or secondary hypertension)
* Normotensive control subjects
* Subjects with aortic stenosis (subgroup "aortic stenosis")
* Participants of Ironman Triathlon competition

Exclusion Criteria:

* Pregnancy
* Systolic blood pressure <90 mmHg
* Allergies to test compounds

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult hypertensive and normotensive subjects who were treated in Tampere University Hospital clinics of internal medicine or cardiology, or visited medical doctors as outpatients at occupational health care providers in the Pirkanmaa Hospital District.
  Patients with primary aldosteronism from all University clinics (Helsinki, Turku, Kuopio, Oulu) in Finland, who were referred to Tampere University Hospital for adrenal vein sampling.
  Patients with acromegalia from all University clinics (Helsinki, Turku, Kuopio, Oulu) in Finland.
  Participants of Ironman Triathlon competition.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2006-05-25 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in haemodynamic variables during the follow-up | baseline, ten years
  Haemodynamic measurements are performed at baseline, and after approximately 10 years of follow-up
Cardiovascular events | ten years of follow-up
  All cardiovascular events during follow-up

SECONDARY OUTCOMES:
Haemodynamic response to head-up tilt and research drugs | 0, 5, 10, 15, 20, 25 and 30 minutes
  Rapid haemodynamic responses are assessed during the same measurement session (the response to head-up tilt and to research drugs salbutamol, nitroglycerin and L-arginine)
Haemodynamic response to bisoprolol or dietary supplements (liquorice, milk casein-derived polypeptides) | baseline and after 2 weeks (liquorice); 3 weeks (bisoprolol), or 12 weeks (polypeptides)
  The change in haemodynamic variables after daily consumption of liquorice (2 weeks); bisoprolol (3 weeks); small milk casein-derived polypeptides (12 weeks)
Haemodynamic changes induced by Ironman competition | Recordings within 2 hours after completion Ironman competition, 12-18 hours later, and within 1-4 before or 4-8 weeks after the competition
  Recordings are performed during normal conditions (training peroid) and after completion of a full-length Ironman competition

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Pörsti, MD, PhD, Principal Investigator — Tampere University
Locations (2):
- Finland (2):
  - Tampere University, Tampere, Southern Finland
  - Tampere University Hospital, Tampere, Southern Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Taurio J, Hautaniemi EJ, Koskela JK, Eraranta A, Hamalainen M, Tikkakoski A, Kettunen JA, Kahonen M, Niemela O, Moilanen E, Mustonen J, Porsti I. The characteristics of elevated blood pressure in abdominal obesity correspond to primary hypertension: a cross-sectional study. BMC Cardiovasc Disord. 2023 Mar 27;23(1):161. doi: 10.1186/s12872-023-03150-w. PMID 36973671
- [Derived] Koskela JK, Tahvanainen A, Tikkakoski AJ, Kangas P, Uitto M, Viik J, Kahonen M, Mustonen J, Porsti I. Resting heart rate predicts cardiac autonomic modulation during passive head-up tilt in subjects without cardiovascular diseases. Scand Cardiovasc J. 2022 Dec;56(1):138-147. doi: 10.1080/14017431.2022.2079713. PMID 35652524
- [Derived] Hamid H, Kurra V, Choudhary MK, Bouquin H, Niemela O, Kahonen MAP, Mustonen JT, Porsti IH, Koskela JK. Plasma uric acid is related to large arterial stiffness but not to other hemodynamic variables: a study in 606 normotensive and never-medicated hypertensive subjects. BMC Cardiovasc Disord. 2021 May 26;21(1):257. doi: 10.1186/s12872-021-02072-9. PMID 34039285
- [Derived] Kokko E, Nevalainen PI, Choudhary MK, Koskela J, Tikkakoski A, Huhtala H, Niemela O, Viukari M, Mustonen J, Matikainen N, Porsti I. Aldosterone-to-renin ratio is related to arterial stiffness when the screening criteria of primary aldosteronism are not met. Sci Rep. 2020 Nov 13;10(1):19804. doi: 10.1038/s41598-020-76718-7. PMID 33188272
- [Derived] Hautaniemi EJ, Tikkakoski AJ, Eraranta A, Kahonen M, Hamalainen E, Turpeinen U, Huhtala H, Mustonen J, Porsti IH. Liquorice ingestion attenuates vasodilatation via exogenous nitric oxide donor but not via beta2-adrenoceptor stimulation. PLoS One. 2019 Oct 18;14(10):e0223654. doi: 10.1371/journal.pone.0223654. eCollection 2019. PMID 31626649
- [Derived] Kangas P, Tahvanainen A, Tikkakoski A, Koskela J, Uitto M, Viik J, Kahonen M, Koobi T, Mustonen J, Porsti I. Increased Cardiac Workload in the Upright Posture in Men: Noninvasive Hemodynamics in Men Versus Women. J Am Heart Assoc. 2016 Jun 21;5(6):e002883. doi: 10.1161/JAHA.115.002883. PMID 27329447
- [Derived] Wilenius M, Tikkakoski AJ, Tahvanainen AM, Haring A, Koskela J, Huhtala H, Kahonen M, Koobi T, Mustonen JT, Porsti IH. Central wave reflection is associated with peripheral arterial resistance in addition to arterial stiffness in subjects without antihypertensive medication. BMC Cardiovasc Disord. 2016 Jun 7;16:131. doi: 10.1186/s12872-016-0303-6. PMID 27266507
- [Derived] Tahvanainen AM, Tikkakoski AJ, Koskela JK, Nordhausen K, Viitala JM, Leskinen MH, Kahonen MA, Koobi T, Uitto MT, Viik J, Mustonen JT, Porsti IH. The type of the functional cardiovascular response to upright posture is associated with arterial stiffness: a cross-sectional study in 470 volunteers. BMC Cardiovasc Disord. 2016 May 23;16:101. doi: 10.1186/s12872-016-0281-8. PMID 27216309
- [Derived] Leskinen MH, Hautaniemi EJ, Tahvanainen AM, Koskela JK, Paallysaho M, Tikkakoski AJ, Kahonen M, Koobi T, Niemela O, Mustonen J, Porsti IH. Daily liquorice consumption for two weeks increases augmentation index and central systolic and diastolic blood pressure. PLoS One. 2014 Aug 25;9(8):e105607. doi: 10.1371/journal.pone.0105607. eCollection 2014. PMID 25153328
- [Derived] Koskela JK, Tahvanainen A, Haring A, Tikkakoski AJ, Ilveskoski E, Viitala J, Leskinen MH, Lehtimaki T, Kahonen MA, Koobi T, Niemela O, Mustonen JT, Porsti IH. Association of resting heart rate with cardiovascular function: a cross-sectional study in 522 Finnish subjects. BMC Cardiovasc Disord. 2013 Nov 15;13:102. doi: 10.1186/1471-2261-13-102. PMID 24237764